CLINICAL TRIAL: NCT02928965
Title: The Benefit of Minocycline on Negative Symptoms in Schizophrenia: Extent and Mechanisms
Acronym: BeneMin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: University of Edinburgh (Other); University of Cambridge (Other); University College, London (Other); University of Birmingham (Other); King's College London (Other); Manchester Mental Health & Social Care Trust (Other Government); Greater Manchester Mental Health NHS Foundation Trust (Other); Northern Care Alliance NHS Foundation Trust (Other); Lancashire Care NHS Foundation Trust (Network); Cambridgeshire and Peterborough NHS Foundation Trust (Other); West London Mental Health NHS Trust (Other); North East London Foundation Trust (Other); Central and North West London NHS Foundation Trust (Other); Camden and Islington NHS Foundation Trust (Unknown); South London and Maudsley NHS Foundation Trust (Other); NHS Lothian (Other Government); NHS Fife (Other Government); NHS Borders (Other Government); University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Bill Deakin, Professor of Psychiatry and Director of Neuroscience Research in the Division of Psychiatry, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EME-09/100/23; 2010-022463-35 (EudraCT Number); 10411 (Other: United Kingdom Clinical Research Network)
Record Dates: First submitted 2016-09-23; First posted 2016-10-10 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2017-10

CONDITIONS: Schizophrenia and Disorders With Psychotic Features
Keywords: psychosis; schizophrenia; negative symptoms; minocycline
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Psychotic Disorders; Schizophrenia; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline (Experimental): Participants will receive capsules containing 100mg of minocycline (modified release), two per day for the first two weeks of the trial and then three per day for the remainder of the 12 month treatment period in addition to antipsychotic drug treatment and other interventions by the responsibel medical officer.
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator): Participants will receive placebo capsules entirely matching minocycline, two per day for the first two weeks of the trial and then three per day for the reminder of the 12 month treatment period in addition to antipsychotic drug treatment and other interventions by the responsibel medical officer.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minocycline — Capsules containing 100mg minocycline (modified release), administered orally by the patient, two per day for the first two weeks and then three per day for the reminder of the 12 month treatment period in addition to standard therapy.
  Other Names: Acnamino MR (modified release)
  Arms: Minocycline
Drug: Placebo — Matching placebo with appearance of over - encapsulated minocycline
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate if minocycline limits the development of negative symptoms in early psychosis and to test via what mechanism of action this change occurs.

DETAILED DESCRIPTION:
Background

Negative symptoms of psychosis do not respond to the traditional therapy with first- or second-generation antipsychotics and are among main causes of a decrease in quality of life observed in individuals suffering from the disorder. Minocycline, a broad-spectrum tetracyclic antibiotic displaying neuroprotective properties has been suggested as a new potential therapy for negative symptoms. In the two previous clinical trials comparing minocycline and placebo, both added to the standard care, patients receiving minocycline showed increased reduction in negative symptoms. Three routes to neuroprotection by minocycline have been identified: neuroprotection against grey matter loss, anti-inflammatory action and stabilisation of glutamate receptors. However, it is not yet certain what the extent of the benefit of minocycline in psychosis is and what its mechanism is. This proposal is for a multi-centre double-blind randomised placebo-controlled clinical trial entitled The Benefit of Minocycline on Negative Symptoms of Psychosis: Extent and Mechanism (BeneMin).

Methods

After providing informed consent, 226 participants in the early phase of psychosis will be randomised to receive either 100 mg modified-release capsules of minocycline or similar capsules with placebo for 12 months in addition to standard care. The participants will be tested for outcome variables before and after the intervention period. The extent of benefit will be tested via clinical outcome measures, namely the Positive and Negative Syndrome Scale score, social and cognitive functioning scores, antipsychotic medication dose equivalent and level of weight gain. The mechanism of action of minocycline will be tested via blood screening for circulating cytokines and magnetic resonance imaging with three-dimensional T1-weighted rapid gradient-echo, proton density T2-weighted dual echo and T2*-weighted gradient echo planar imaging with N-back task and resting state. Eight research centres in the United Kingdom (UK) and 15 National Health Service Trusts and Health Boards will be involved in recruiting participants, performing the study and analysing the data.

ELIGIBILITY:
Inclusion Criteria:

* Meeting DSM-IV criteria for schizophrenia, schizophreniform or schizo-affective psychosis as assessed by the research team
* In an episode as defined by the presence of positive symptoms measured by Positive and Negative Syndrome Scale with a score higher than two in items 1,2,3 or 6 in the Positive scale
* In contact with early intervention community or in-patient service
* Within 5 years of first diagnosis
* Intelligence quotient (IQ) greater than 70
* Participants and their partners must be willing to use effective birth control throughout the study and seven days after stopping trial medication. Females should have a negative pregnancy test
* Able to understand and willing to give written informed consent
* Fluent in English

Exclusion Criteria:

* Current substance misuse diagnosis that in the opinion of the investigator may interfere with the study
* Patients who, in the investigator's judgement pose a current serious suicidal or violence risk
* Use of tetracycline antibiotics within 2 months of the randomisation visit or history of sensitivity or intolerance for this type of antibiotics
* History of Systemic Lupus Erythematosis (SLE) or a history of SLE in a first-degree relative
* Use of any investigational drug within a month of randomisation visit
* Relevant current or past hematologic, hepatic, renal, neurological or other medical disorder in the opinion of the principal investigator (PI) or the responsible medical officer (RMO) may interfere with the trial
* Taking medical treatments that could seriously interact with minocycline as described in the summary of product characteristics (SPC) and judged by the PI or the RMO
* Clinically significant deviation from the reference range in clinical laboratory test results as judged by the investigator
* Previous randomisation in the present study
* Pregnant or breastfeeding
* Meeting MRI exclusion criteria as defined by local scanning centres

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 207 (Actual)
Dates: Start 2013-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Severity of negative symptoms of psychosis | twelve months
  Measured by Negative symptoms scale in the Positive and Negative Syndrome Scale

SECONDARY OUTCOMES:
Change in body weight | Twelve months
  Measuring weight gain in kilograms, a side effect of standard anti-psychotic medication therapy
Positive symptoms of psychosis | twelve months
  Measured by the Positive symptoms scale in the Positive and Negative Syndrome Scales
General social and psychological functioning | twelve months
  Measured by Global Assessment of Functioning from DSM-IV
Intelligence | twelve months
  Measured by Wechsler Adult Intelligence Scale for patients with schizophrenia
Anti-psychotic medication dose | twelve months
  Measured in chlorpromazine equivalent units
Verbal learning | 12 months
  Auditory-Verbal Learning Task
Social and Occupational functioning | 12 months
  Score on Social Functioning Scale

OTHER OUTCOMES:
Change in medial prefrontal grey matter volume (primary biomarker outcome) | twelve months
  Change Measured by T1-weighted magnetic resonance imaging (MRI)
Circulating interleukin (IL-6) concentration (primary biomarker outcome) | twelve months
  Measured by blood cytokine screen test
Dorsolateral-prefrontal cortex blood oxygen level dependent response during working memory task (primary biomarker outcome) | twelve months
  Measured by functional magnetic resonance imaging during N-back task
Pattern of total and regional grey matter volumes (secondary biomarker outcome) | twelve months
  Measured by T1-weighted magnetic resonance imaging
Multivariate pattern of circulating cytokine concentrations (secondary biomarker outcome) | twelve months
  Measured by blood cytokine screen test
Distribution of Hurst exponent (brain functional connectivity measure; secondary biomarker outcome) | twelve months
  Measured by functional magnetic resonance imaging during resting state
Verbal fluency | 12 months
  Verbal fluency, words per minute beginning with F, A and S
Working memory | 12 months
  Performance on the N-back task during scanning

CONTACTS AND LOCATIONS:
Overall Officials: Bill Deakin, Professor, Principal Investigator — University of Manchester

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymised database will be made available in 2018. Basic demographics, Primary clinical and mechanistic outcome measures. Treatment allocation code
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: January 2019
Access Criteria: Academic researcher, clear analysis plan, publication plan Agreement of Chief investigator